CLINICAL TRIAL: NCT04731987
Title: Orange Juice, Hesperidin and Their Role in Vascular Health Benefit: a Human Double Blind, Randomized, Controlled, Cross Over Study
Brief Title: Orange Juice, Hesperidin and Their Role in Vascular Health Benefit
Acronym: HESPER-HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UMR 1019, Unité de Nutrition Humaine, INRAE, Auvergne-Rhône Alpes Center (Unknown); Department of Beverage Research, Chair of analysis and technology of plant-based foods, Geisenheim University (Unknown); European Fruit Juice Association (AIJN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RBHP 2020 PICKERING 2
Record Dates: First submitted 2021-01-22; First posted 2021-02-01 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Syndrome; Vascular Compliance; Predisposition to Cardiovascular Disease
Keywords: Cardiovascular disease prevention; Endothelial dysfunction; Orange juice; Flavanone; Hesperidin; Nutrition Assessment; Nutritional Physiological Phenomena
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: drinks kits will be labelled and packaged according to the pre-established randomization plane by the pharmacy department of University Hospital of Clermont-Ferrand, France. Kits will be distributed in a blind fashion for each cross over period on the basis of the randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Orange juice (A) (Experimental): 42 subjects between 40 and 65 years old with predisposition to cardiovascular disease will consume daily 330 ml of orange juice naturally rich in hesperidin (drink A) during 6 weeks
  Interventions: Behavioral: Beverage consumption
- Control beverage (B) (Placebo Comparator): 42 subjects between 40 and 65 years old with predisposition to cardiovascular disease will consume daily 330 ml of control beverage (drink B)- a soft drink with sugar concentration identical to drink A - during 6 weeks
  Interventions: Behavioral: Beverage consumption
- Control beverage supplemented with hesperidin formulation (B+HESP) (Experimental): 42 subjects between 40 and 65 years old with predisposition to cardiovascular disease will consume daily 330 ml of control beverage (identical to drink B but supplemented with hesperidin to reach level of drink A) during 6 weeks
  Interventions: Behavioral: Beverage consumption

INTERVENTIONS:
Behavioral: Beverage consumption — Volunteers will consume, in random order, daily 330 ml of 1 experimental beverage per period (Orange Juice, Control Beverage, Control Beverage supplemented with hesperidin) for 6 weeks in each period.
  At the beginning and the end of each period, exploration will be conducted at fasted state and at post-prandial state after the administration of a high-fat high-sugar meal.

SUMMARY:
Although epidemiological studies have associated the consumption of sugary beverages with adverse health effects, experimental studies have demonstrated that the metabolic response of the human body to fruit juice as compared to artificial beverages is substantially different. Fruit juices do not just provide sugars and related calories, but they are rich sources of bioactive compounds especially of flavonoids. Flavanones constitute a class of flavonoids that are specifically and abundantly found in citrus fruits, with hesperidin being the major compound in orange. From prospective cohort studies, higher intakes of flavanones are associated with a lower incidence of mortality by cardiovascular disease (CVD). This relation is supported by results from a number of animal studies demonstrating a slowdown in atherosclerosis development and vascular protective effects in dietary interventions with flavanones. Randomized, controlled clinical trials to corroborate the suggested vasculo-protective effects of orange juice presumably mediated by the flavanones are scarce and available data do not allow to draw firm conclusions about their efficacy. To fill this gap, the "HESPER-HEALTH study" conducted in humans will assess the vascular protective effects of 100% orange juice consumption and evaluate the contribution of hesperidin in these effects.

DETAILED DESCRIPTION:
This human dietary intervention study is a double blind, randomized, placebo controlled, cross over trial with 3 arms, carried out on subjects with predisposition to cardiovascular diseases (CVD) based on age and overweight. This study aims to demonstrate the vascular protective effects (with Flow Mediated Dilatation (FMD) as main criteria) of the consumption of a flavanone rich orange juice or of orange flavanones by comparison with a control sugary drink alone.

The 42 recruited participants will receive the 3 drinks in a random order. For each subject, the study is divided into 3 identical experimental periods of 45 days (period 1,2,3): including 3 days prior to the beginning of the product intake, during which specific dietary guidelines, samplings and measures will be asked to be performed at home followed by a 6 weeks period of consumption of each of the 3 beverages). A period of 4 to 6 weeks of wash-out is planned between each experimental period.

To summarize: Visit 1 (D-14) = inclusion, Visit 2 (D1: baseline) to 3 (D42) = period 1, Visit 3 (D42) to 4 (D70) = wash out 1, Visit 4 (D70) to 5 (D111) = period 2, Visit 5 (D111) to 6 (D139) = wash out 2, Visit 6 (D139) to 7 (D180) = period 3. The wash-out periods (minimum duration: 4 weeks) may be extended until 6 weeks for the convenience of participants.

The protocol includes a total of 7 visits to PIC/CIC Inserm 1405 of the Clermont-Fd University Hospital.

The total duration of the study will be between 28 and 34 weeks

ELIGIBILITY:
Inclusion Criteria:

* Man or post-menopausal woman ;
* 40-65 years old (inclusive) ;
* Body Mass Index (BMI)≤ 30 ;
* Waist circumference ≥80 cm for women, and ≥94 cm for men ;
* Weight > 46 kg
* Normal biological balance sheet or considered normal by the investigator
* No aversion or intolerance to citrus foods ;
* Accept to limit their total intake of flavonoid rich beverages (tea, coffee, cocoa, wine, fruit juice) to 250 mL/day ;
* Ability to give informed consent to participate in research ;
* Willingness to accept randomization and undergo the testing and intervention procedures and deliver stool, blood and urine samples for testing ;
* Affiliation to Social Security.

Exclusion Criteria:

* Treated pre-diabetic or diabetic ;
* Treated for hypertension ;
* Use of statins or other medications for lowering cholesterol ;
* Treated with antibiotics, antifungals, probiotics or prebiotics in the 3 months before the enrolment ;
* Menopausal hormone replacement therapy ;
* Diagnosed gastrointestinal illness in the judgement of the investigator ;
* Any serious medical condition that precludes safe participation in the study, such as coronary artery disease, peripheral vascular disease, stroke, congestive heart failure, chronic obstructive pulmonary disease, insulin-dependent diabetes, psychiatric disease, renal disease, liver disease, active cancer and anemia ;
* History of eating disorders such as bulimia nervosa, anorexia nervosa and severe binge eating disorder in the last 5 years ;
* Digestive disorders with diarrhea during the 3 months preceding the beginning of the study ;
* Self-declared vegetarian, vegetalian, vegan ;
* History of substance abuse or alcohol abuse ;
* Involvement in a weight loss intervention program (including anti-obesity medication) within the past 3 months or who have had bariatric surgery ;
* Current smokers (within the last 30 days) ;
* Use of dietary supplements (vitamins, antioxidants) currently or in the past one month ;
* Strenuous exercise greater than 6 hours per week ;
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol ;
* Subjects involved in another clinical trial or being in the exclusion period of another study or having received a total compensation greater than 4,500 euros over the 12 months preceding the start of the trial ;
* Subject benefiting from a legal protection measure (curatorship, guardianship, safeguard of justice) ;
* Refusal to participate.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Brachial artery Flow Mediated Dilation (FMD) | Day 1
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery in fasted state
Brachial artery Flow Mediated Dilation (FMD) | Day 42
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery in fasted state
Brachial artery Flow Mediated Dilation (FMD) | Day 70
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery in fasted state
Brachial artery Flow Mediated Dilation (FMD) | Day 111
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery in fasted state
Brachial artery Flow Mediated Dilation (FMD) | Day 139
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery in fasted state
Brachial artery Flow Mediated Dilation (FMD) | Day 180
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery in fasted state

SECONDARY OUTCOMES:
Sex | Day -14
  Participant sex (man/women) will be requested.
Age | Day 34
  Participant age (years) will be requested.
Basal Systolic Blood Pressure | Day -14
  Blood pressure measure (mm Hg) with monitor.
Basal Heart Rate | Day -14
  Heart rate measure (beat/min) with monitor.
D-3 visit systolic Blood Pressure (BP) | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Self-monitored blood pressure (mmHg) at home with tensiometer, at home the morning, 3 days before the visit, in fasted state.
D-3 visit diastolic BP | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Self-monitored blood pressure (mmHg) at home with tensiometer, at home the morning, 3 days before the visit, in fasted state.
D-3 visit Heart Rate | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Self-monitored heart rate (beat/min) at home with tensiometer,at home the morning, 3 days before the visit, in fasted state.
FMD post prandial endothelial response 3h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Assessment of the postprandial endothelial response to a challenge meal (900kcal, fresh cream, sucrose and milk proteins) by measuring FMD (percent) using ultrasound technique, 3h after intake of the full daily dose of study products concomitantly with challenge meal.
FMD post prandial endothelial response 6h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Assessment of the postprandial endothelial response to a challenge meal by measuring FMD (percent) using ultrasound technique, 6h after intake of the full daily dose of study products concomitantly with challenge meal.
Arterial compliance assessment | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Noninvasive measure with Sphygmocor (AtCor Medical Pty. Ltd) of pulse transit time between carotid artery and femoral artery. The carotid-femoral Pulse Wave Velocity (PWV) (m/sec) is an established index of arterial stiffness,in fasted state.
Rest flow by Flowmetry Laser Doppler (FLD) in fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the rest flow using laser-Doppler system at the level of the skin of the hand, in fasted state
Occlusion area by FLD in fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the occlusion area using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement) in fasted state
Hyperaemia area by FLD in fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the hyperaemia area using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement) in fasted state
Hyperaemia area / occlusion area ratio by FLD in fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the ratio hyperaemia area / occlusion area determined by FLD.
Maximal flow by FLD in fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the maximal flow using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), in fasted state
Hyperaemia half time by FLD in fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the hyperaemia half time using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), in fasted state
Rest flow by FLD 3h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the rest flow using laser-Doppler system at the level of the skin of the hand,3h after intake of the full daily dose of study products concomitantly with challenge meal
Occlusion area by FLD 3h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the occlusion area using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), 3h after intake of the full daily dose of study products concomitantly with challenge meal
Hyperaemia area by FLD 3h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the hyperaemia area using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), 3h after intake of the full daily dose of study products concomitantly with challenge meal
Hyperaemia area / occlusion area ratio by FLD 3h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the ratio hyperaemia area/ occlusion area determined by FLD, 3h after intake of the full daily dose of study products concomitantly with challenge meal
Maximal flow by FLD 3h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the maximal flow using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), 3h after intake of the full daily dose of study products concomitantly with challenge meal
Hyperaemia half time by FLD 3h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the hyperaemia half time using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), 3h after intake of the full daily dose of study products concomitantly with challenge meal
Rest flow by FLD 6h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the rest flow using laser-Doppler system at the level of the skin of the hand, 6h after intake of the full daily dose of study products concomitantly with challenge meal
Occlusion area by FLD 6h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the occlusion area using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), 6h after intake of the full daily dose of study products concomitantly with challenge meal
Hyperaemia area by FLD 6h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the hyperaemia area using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), 6h after intake of the full daily dose of study products concomitantly with challenge meal
Hyperaemia area / occlusion area ratio by FLD 6h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the ratio hyperaemia area / occlusion area ratio determined by FLD, 6h after intake of the full daily dose of study products concomitantly with challenge meal
Maximal flow by FLD 6h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the maximal flow using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), 6h after intake of the full daily dose of study products concomitantly with challenge meal
Hyperaemia half time by FLD 6h after a challenge meal | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the hyperaemia half time using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement), 6h after intake of the full daily dose of study products concomitantly with challenge meal
Hesperetin concentration in 24h urine | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of hesperetin in urine (nM) will be measured.
Hesperetin concentration in plasma on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of hesperetin in plasma (nM) will be measured.
Hesperetin catabolites concentration in plasma on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of hesperetin microbial catabolites in plasma (nM) will be measured, on fasted state
Hesperetin concentration in plasma on 3h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of hesperetin in plasma (mM) will be measured, in post prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Hesperetin catabolites concentration in plasma on 3h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of hesperetin microbial catabolites in plasma (mM) will be measured, in post prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Hesperetin concentration in plasma on 6h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of hesperetin in plasma (mM) will be measured, in post prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Hesperetin catabolites concentration in plasma on 6h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of hesperetin microbial catabolites in plasma (mM) will be measured, in post prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Naringenin concentration in 24h urine | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of naringenin in urine (nM) will be measured.
Naringenin catabolites concentration in 24h urine | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of naringenin microbial catabolites in urine (nM) will be measured.
Naringenin concentration in plasma on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of naringenin in plasma (nM) will be measured, on fasted state
Naringenin catabolites concentration in plasma on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of naringenin microbial catabolites in plasma (nM) will be measured, on fasted state
Naringenin concentration in plasma on 3h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of naringenin in plasma (mM) will be measured, in post prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Naringenin catabolites concentration in plasma on 3h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of naringenin microbial catabolites in plasma (mM) will be measured, in post prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Naringenin concentration in plasma on 6h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of naringenin in plasma (mM) will be measure, in post prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Naringenin catabolites concentration in plasma on 6h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of naringenin microbial catabolites in plasma (mM) will be measured, in post prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Flavanone concentration in 24h urine | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of flavanone in urine (nM) will be measured.
Flavanone catabolites concentration in 24h urine | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of flavanone microbial catabolites in urine (nM) will be measured.
Flavanone concentration in plasma on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of flavanone in plasma (nM) will be measured, on fasted state.
Flavanone catabolites concentration in plasma on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of flavanone microbial catabolites in plasma (nM) will be measured, on fasted state
Flavanone concentration in plasma on 3h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of flavanone in plasma (mM) will be measured, in post prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Flavanone catabolites concentration in plasma on 3h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of flavanone microbial catabolites in plasma (mM) will be measured,in post prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Flavanone concentration in plasma on 6h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of flavanone in urine (nM) will be measured, in post prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Flavanone catabolites concentration in plasma on 6h post prandial test | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Concentration of flavanone microbial catabolites in plasma (mM) will be measured, in post prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Plasma nitrites dosage | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of nitrite plasma concentration (nM) (a biomarker of endothelial activation), on fasted state
Plasma nitroso-thiols dosage | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of nitroso-thiols plasma concentration (nM) (a biomarker of endothelial activation), on fasted state
Plasma Inter-Cellular Adhesion Molecules (ICAM) dosage on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of ICAM plasma concentration (ng/ml) (a biomarker of endothelial activation), on fasted state
Plasma ICAM dosage on 6h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of ICAM plasma concentration (ng/ml) (a biomarker of endothelial activation), on 6h post prandial state
Plasma Vascular-CAM (VCAM) dosage on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of VCAM plasma concentration (ng/ml) (a biomarker of endothelial activation), on fasted state
Plasma VCAM dosage on 6h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of VCAM plasma concentration (ng/ml) (a biomarker of endothelial activation), on 6h post prandial state
Plasma e-selectin dosage on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of e-selectin plasma concentration (ng/ml) (a biomarker of endothelial activation), on fasted state
Plasma e-selectin dosage on 6h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of e-selectin plasma concentration (ng/ml) (a biomarker of endothelial activation), on 6h post prandial state
Plasma Extracellular Vesicles analyses (EVs) on fasted state | Day 42, Day 111, Day 180
  EVs (a biomarker of endothelial activation) will be isolated from platelet-poor plasma samples and analyzed, on fasted state
EVs analyses on 3h post prandial state | Day 42, Day 111, Day 180
  EVs (a biomarker of endothelial activation) will be isolated from platelet-poor plasma samples and analyzed, on post prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Plasma oxylipins identification on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of oxylipins present in plasma (a biomarker of inflammation and oxidative stress) using a method of profiling, on fasted state
Plasma oxylipin concentration on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of oxylipin plasma concentration (a biomarker of inflammation and oxidative stress), on fasted state
Plasma oxylipins identification on 6h post prandial state | Day 42, Day 111, Day 180
  Determination of oxylipins present in plasma (a biomarker of inflammation and oxidative stress) using a method of profiling, on post-prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Plasma oxylipin concentration on 6h post prandial state | Day 42, Day 111, Day 180
  Determination of oxylipin plasma concentration (a biomarker of inflammation and oxidative stress), on post-prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Plasma Interleukin 6 (IL-6) dosage | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of IL-6 plasma concentration (pg/ml) (a biomarker of inflammation and oxidative stress), on fasted state
Plasma Tumor Necrosis Factor α (TNFα) dosage | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of TNFα plasma concentration (pg/ml) (a biomarker of inflammation and oxidative stress), on fasted state
Plasma high-sensitivity C-reactive protein (hs-CRP) dosage | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of hs-CRP plasma concentration (mg/L) (a biomarker of inflammation and oxidative stress), on fasted state
Plasma glucose dosage on fasted state | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of glucose plasma concentration (mM) (a metabolic parameter), on fasted state
Plasma glucose dosage on 3h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of glucose plasma concentration (mM) (a metabolic parameter), on post-prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Plasma glucose dosage on 6h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of glucose plasma concentration (mM) (a metabolic parameter), on post-prandial state 6h after the concomitant consumption of the study drink and challenge meal.
-Plasma Triacylglycerol (TAG) dosage on fasted state | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of TAG plasma concentration (g/L) (a metabolic parameter), on fasted state
Plasma TAG dosage on 3h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of TAG plasma concentration (g/L) (a metabolic parameter), on post-prandial state 3h after the concomitant consumption of the study drink and challenge meal, on post-prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Plasma TAG dosage on 6h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of TAG plasma concentration (g/L) (a metabolic parameter), on post-prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Plasma uric acid dosage on fasted state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of uric acid plasma concentration (mM) (a metabolic parameter) method, on fasted state
Plasma uric acid on 3h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of uric acid plasma concentration (mM) (metabolic parameter), on post-prandial state 3h after the concomitant consumption of the study drink and challenge meal.
Plasma uric acid on 6h post prandial state | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of uric acid plasma concentration (mM) (metabolic parameter) will be determined, on post-prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Plasma total cholesterol dosage | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of total cholesterol plasma concentration (mM) (a metabolic parameter), on fasted state
Plasma High Density Lipoprotein cholesterol (HDL-chol) dosage | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of HDL-chol plasma concentration (mM) (a metabolic parameter), on fasted state
Plasma High Density Lipoprotein cholesterol (LDL-chol) calculation | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of LDL-chol plasma concentration (mM) (metabolic parameter), on fasted state
Plasma Total Fatty Acids (FA) dosage | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of total FA plasma concentration (mM) (a metabolic parameter), on fasted state
Serum Insulin dosage | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Determination of insulin serum concentration (mU/L or pM) (a metabolic parameter), on fasted state
Weight measure | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  the body weight (kg) will be recorded with a bathroom scale, on fasted state
Height measure | Day -14
  the body height (cm) will be measured with a stadiometer.
Body Mass Index (BMI) calculation | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  the BMI (kg/m²) will be calculated, on fasted state
Waist circumference measure | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  the waist circumference (cm) will be recorded with a measuring tape, on fasted state
Fat mass ratio determination | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  The percentage of fat mass (percent) (body composition) will be determined on each participant using a multi-frequency bioelectrical Impedance Analyzer, on fasted state
Lean mass ratio determination | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  The percentage of lean mass (percent) (body composition) will be determined on each participant using a multi-frequency bioelectrical Impedance Analyzer, on fasted state
Water mass ratio determination | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  The percentage of water (percent) (body composition) will be determined using a multi-frequency bioelectrical Impedance Analyzer, on fasted state
RNA profiling on fasted state | Day 42, Day 111, Day 180
  Nutrigenomic analysis will be performed from total Ribo Nucleic Acid (RNA) isolated blood collected in PAXgene Blood RNA Tube. The isolated RNA will be used to perform microarray analyses that allow identification of expression of all genes of the genome, on fasted state
RNA profiling on 6h post prandial state | Day 42, Day 111, Day 180
  Analysis will be performed from total RNA isolated blood collected in PAXgene Blood RNA Tube. The isolated RNA will be used to perform microarray analyses that allow identification of expression of all genes of the genome, on post-prandial state 6h after the concomitant consumption of the study drink and challenge meal.
Gut microbiota profiling | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Identification of the microbiota composition of feces samples (collected by subjects) by performing a genetic sequencing analysis of bacterial DNA.
Plasma carotenoids dosage | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Carotenoids will be quantitated from plasma (nM), on fasted state
Plasma vitamine C dosage | Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Vitamin C status will be quantified in deproteinized plasma (mg/L), on fasted state
Treatment compliance | Day 42, Day 111, Day 180
  Treatment compliance (percent) will be determined using counting of empty orange drinks brought back by volunteers after the consumption periods
Polyphenol intake | Day 1, Day 42, Day 111, Day 180
  Polyphenol intake (ml/day) in basal and during treatment consumption periods will be determined by a dietician using food report completed by volunteers.
Low-polyphenol diet compliance | Day 1, Day 42, Day 111, Day 180
  Respect (y/n) of a low-polyphenol diet in basal (between Visit 1 - Visit 2) and during treatment consumption periods (between Visit 2 - Visit 3, Visit 4 - Visit 5, Visit 6 - Visit 7) will be determined by a dietician using 3 days food reports completed by volunteers.
Calorie intake | Day 1, Day 42, Day 111, Day 180
  Calorie (kcal/day) intake in basal and during treatment consumption periods will be determined by a dietician using food report completed by volunteers.
Protein intake | Day 1, Day 42, Day 111, Day 180
  Protein (g/day) intake in basal and during treatment consumption periods will be determined by a dietician using food report completed by volunteers.
Lipid intake | Day 1, Day 42, Day 111, Day 180
  Lipid intake (g/day) in basal and during treatment consumption periods will be determined by a dietician using food report completed by volunteers.
Carbohydrate intake | Day 1, Day 42, Day 111, Day 180
  Carbohydrate intake (g/day) in basal and during treatment consumption periods will be determined by a dietician using food report completed by volunteers.
Diet division of protein/lipid/carbohydrate intakes | Day 1, Day 42, Day 111, Day 180
  The overall distribution of the protein/lipid/carbohydrate food intakes (%) will be determined by a dietician using food report completed by volunteers.
Diet stability | Day 180
  Diet stability (y/n) in terms of polyphenols, calories, proteins, carbohydrates and lipids intakes during the whole study will be determined by a dietician using the 4 food reports completed by volunteers.
Biobank for food metabolome | Day -14, Day 1, Day 42, Day 70, Day 111, Day 139, Day 180
  Urine samples will be stored for further assessment of food metabolome to potentially identify new bioactive compounds present in the juice that could contribute to the biological response after orange juice/HESP intake.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont Ferrand, Clermont-Ferrand, AURA, France

REFERENCES:
- [Derived] Verny MA, Milenkovic D, Macian N, Pereira B, Evrard R, Gilcher C, Steingass CB, Mosoni P, Gladine C, Monfoulet LE, Schweiggert R, Pickering G, Morand C. Evaluating the role of orange juice, HESPERidin in vascular HEALTH benefits (HESPER-HEALTH study): protocol for a randomised controlled trial. BMJ Open. 2021 Nov 30;11(11):e053321. doi: 10.1136/bmjopen-2021-053321. PMID 34848522